CLINICAL TRIAL: NCT01585103
Title: Cytosponge Protocol
Brief Title: Cytosponge Protocol IRB 11-006429
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device was recalled by company
Sponsor: Mayo Clinic (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Jeffrey A Alexander, Prinicipal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-006429
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2022-05-18 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Cytosponge/ brushing (Experimental): Subjects with eosinophilic esophagitis undergoing clinically indicated endoscopy and biopsy either for initial diagnosis or for monitoring the activity of their disease will be asked to swallow the cytosponge two hours prior to endoscopy.
  Interventions: Device: Cytosponge

INTERVENTIONS:
Device: Cytosponge — An ingestible gelatin capsule containing a compressed mesh attached to a string. The capsule is swallowed and once in the stomach, the gelatin dissolves and a spherical mesh of 3 cm diameter is released. The mesh is withdrawn through the mouth by the attached string and a cytologic specimen is collected.

SUMMARY:
This study is being done to collect data on the potential use of the cytosponge as non-invasive tool in evaluating patients with eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18 and 65 with eosinophilic esophagitis including lactating or pregnant women undergoing clinically indicated endoscopy and esophageal biopsy.

Exclusion Criteria:

* Patients for whom clinically indicated endoscopy is not safe. Patients who have small caliber esophagus, an esophageal stricture that will not permit passage of the gelatin capsule or are unable to swallow the capsule.
* Vulnerable populations, such as those with diminished mental acuity, will be excluded.
* Patients with known Lidocaine/Acetylcysteine allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Alexander, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katzka DA, Smyrk TC, Alexander JA, Geno DM, Beitia RA, Chang AO, Shaheen NJ, Fitzgerald RC, Dellon ES. Accuracy and Safety of the Cytosponge for Assessing Histologic Activity in Eosinophilic Esophagitis: A Two-Center Study. Am J Gastroenterol. 2017 Oct;112(10):1538-1544. doi: 10.1038/ajg.2017.244. Epub 2017 Aug 15. PMID 28809387
- [Derived] Katzka DA, Geno DM, Ravi A, Smyrk TC, Lao-Sirieix P, Miremadi A, Debiram I, O'Donovan M, Kita H, Kephart GM, Kryzer LA, Camilleri M, Alexander JA, Fitzgerald RC. Accuracy, safety, and tolerability of tissue collection by Cytosponge vs endoscopy for evaluation of eosinophilic esophagitis. Clin Gastroenterol Hepatol. 2015 Jan;13(1):77-83.e2. doi: 10.1016/j.cgh.2014.06.026. Epub 2014 Jul 3. PMID 24997328
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cytosponge/ Brushing
Started | 86
Completed | 80
Not Completed | 6
Not completed — Unable to swallow Cytosponge | 6

BASELINE CHARACTERISTICS:
Arm/Group | Cytosponge/ Brushing
Number analyzed (Participants) | 86
Age, Continuous [Median (Full Range); unit: years] | 42 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Percent Specificity of the Cytosponge
Description: Percent specificity of Cytosponge ability to detect Eosinophilic Esophagitis when compared to upper endoscopy and biopsies/swab testing. Cytology specimens will be reviewed by one pathologist who will read them blindly without knowledge of the results of the biopsy specimens. To calculate specificity: 100% the number of true negatives divided by the sum of the number of true negatives plus the number of false positives.
Time Frame: Baseline
Measure: Number; unit: percentage of samples
Arm/Group | Cytosponge/ Brushing
Number analyzed (Participants) | 80
percentage of samples | 86

2. Primary Outcome: Percent Sensitivity of the Cytosponge
Description: Percent sensitivity of Cytosponge ability to detect Eosinophilic Esophagitis when compared to upper endoscopy and biopsies/swab testing. Cytology specimens will be reviewed by one pathologist who will read them blindly without knowledge of the results of the biopsy specimens. To calculate sensitivity: 100% the number of true positives divided by the sum of the number of true positives plus the number of false negatives
Time Frame: Baseline
Measure: Number; unit: percentage of samples
Arm/Group | Cytosponge/ Brushing
Number analyzed (Participants) | 80
percentage of samples | 75

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to after upper endoscopy for a total of approximately 3 hours on all participants.
Arm/Group | Cytosponge/ Brushing
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 0/86
Other Adverse Events (participants affected / at risk) | 2/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cytosponge/ Brushing (N=86)
Mucosal Tear (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Received a medical device recall for the Cytosponge cell collection device from the manufacturer and study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT01585103/Prot_000.pdf